CLINICAL TRIAL: NCT01704976
Title: Effects of Whole Body Vibration With Stochastic Resonance and Dance Therapy in the Elderly: Effects on Physical Functional Performance
Brief Title: SR-WBV Training for Frail Elderly in the Skilling up Stage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bern University of Applied Sciences (Other)
Responsible Party: Principal Investigator, Slavko Rogan, PTMsc, Bern University of Applied Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MSc-study (Biel)
Record Dates: First submitted 2012-10-07; First posted 2012-10-12 (Estimated); Results first posted 2014-12-24 (Estimated); Last update posted 2019-02-12 (Actual); Status verified 2019-01

CONDITIONS: Poor Performance Status; Muscle Weakness
MeSH Terms: conditions — Muscle Weakness

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): T0 - intervention over 4 weeks with stochastic resonance whole-body vibration (SR-WBV) (5 Hz, noise 4) - T1
  Interventions: Device: SR-WBV
- Sham group (Sham Comparator): T0 - intervention over 4 weeks with stochastic resonance whole-body vibration (SR-WBV) (1 Hz, noise 1) - T1
  Interventions: Device: SR-WBV

INTERVENTIONS:
Device: SR-WBV — Participants will undergo a training program set over four weeks, three times a week with 3 to 6 Hz, Noise 4.
  Other Names: SRT Zeptor® med plus Noise (Swiss Frei AG, Switzerland); Intervention-Group
  Arms: Intervention
Device: SR-WBV — Participants will undergo a training program set over four weeks three times a week with 1 Hz, Noise 1.
  Other Names: SRT Zeptor® med plus Noise (Swiss Frei AG, Switzerland
  Arms: Sham group

SUMMARY:
This randomized controlled study aims to examine long term effects in the skilling up phase over 4 weeks on physical functional performance and strength of mechanical SR-WBV and dance therapy intervention in a frail elderly population.

DETAILED DESCRIPTION:
This study is based on the guideline of falls management exercise programs (FaME; from Skelton and Dinan).

The goals:

Skilling up: improvement in neuromuscular control, postural control and strengthening of large muscle groups of the lower extremity.

Training Gain: improvement of functional abilities. Maintaining the Gains: muscle growth, improvement of bone density and multi-sensory exercises.

First, a pilot study was conducted with untrained elderly ("Effects of stochastic resonance therapy on postural control in the elderly population" (KEK Bern: No.228/09, Clinical Trial Registry: NCT01045746). Following, a second pilot study was conducted with frail elderly (Application of Whole-body Vibration With Stochastic Resonance in Frail Elderly: The Effects on Postural Control Clinical Trial Registry:NCT01543243).

It was found that the selected chosen form of recruitment (presentation and advertisement) and the measurements methods are suitable for untrained elderly. But for frail elderly the chosen form of recruitment and the measurement methods are not sufficient.

For this study, measurement parameters for functional performance and strength will be used.

Goals of the study in the skilling up phase:

1. Feasibility
2. Study the effect on physical functional performance
3. Study the effects on muscle strength.

The participants will be recruited in Canton Bern - Swizerland and will be randomly allocated to an intervention group or sham group.

ELIGIBILITY:
Inclusion Criteria:

* RAI (Resident Assessment Instrument) >0
* live in canton Bern
* in terms of training load be resistant.

Exclusion Criteria:

* acut joint disease, acut thrombosis, acute fractures, acute infections, acute tissue damage, or acute -- surgical scars
* seniors with prosthesis.
* alcoholic
* acute joint disease, activated osteoarthritis, rheumatoid arthritis, acute lower limb
* acute inflammation or infection tumors
* fresh surgical wounds
* severe migraine
* epilepsy
* acute severe pain

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 27 (Actual)
Dates: Start 2012-09; Primary Completion 2014-07 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rogan Slavko, MSc, Study Chair — Bern University of Applied Science, Department WGS; Radlinger Lorenz, PhD, Study Director — Bern University of Applied Science, Department WGS; Baur Heiner, PhD, Principal Investigator — Bern University of Applied Sciences; Jessica Kessler, MSc, Study Chair — BUAS
Locations (1):
- Slavko Rogan, Bern, Switzerland

REFERENCES:
- [Derived] Kessler J, Radlinger L, Baur H, Rogan S. Effect of stochastic resonance whole body vibration on functional performance in the frail elderly: A pilot study. Arch Gerontol Geriatr. 2014 Sep-Oct;59(2):305-11. doi: 10.1016/j.archger.2014.06.005. Epub 2014 Jul 9. PMID 25042993

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: T0 - intervention 4 weeks - T1
  Stochastic resonance whole-body vibration I: Participants will undergo a training program set over four weeks, three times a week with 3 to 6 Hz, Noise 4.
- Sham: T0- Intervention 4 weeks- T1
  Stochastic resonance whole-body vibration II: Participants will undergo a training program set over four weeks three times a week with 1 Hz, Noise 1.
Period: Overall Study
Arm/Group | Intervention | Sham
Started | 14 | 13
Completed | 13 (One participant completed < 11 SR-WBV sessions and was excluded from the statistical analysis) | 11 (2 participants completed < 11 SR-WBV sessions, they were excluded from statistical analysis)
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Sham | Total
Number analyzed (Participants) | 13 | 11 | 24
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 90.7 (7.5) | 83.8 (9.3) | 87.3 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 6 | 4 | 10
Total sum score of the Short Physical Performance Battery Test [Median (Inter-Quartile Range); unit: sum of points] — "Short physical performance battery (SPBB): The SPBB examines three areas of lower extremity function:
  1. standing balance (semi-tandem stand, side-by-side stand, full tandem stand),
  2. walking speed and
  3. ability to stand from a chair. These areas represent essential tasks important for independent living. The scores range from 0 (worst performance) to 12 (best performance). SPPB 0-6 is "Poor performance"; SPPB 7-9 is "Intermediate performance; SPPB 10-12 is "High Performance.".
  sum of points | 3 [2 to 4.5] | 4 [2 to 6] | 3 [2 to 5]

OUTCOME MEASURES:

1. Primary Outcome: Physical Functional Performance
Description: Short physical performance battery (SPBB): The SPBB examines 3 areas of lower extremity function: standing balance (semi-tandem stand, side-by-side stand, full tandem stand), usual walking speed and ability to stand from a chair. These areas represent essential tasks important for independent living.
  The scores range from 0 (worst performance) to 12 (best performance). SPPB 0-6 is "Poor performance"; SPPB 7-9 is "Intermediate performance; SPPB 10-12 is "High Performance".
Time Frame: after 4 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Intervention | Sham
Number analyzed (Participants) | 13 | 11
units on a scale
  Pre-intervention | 3 [2 to 4.5] | 4 [2 to 6]
  Post-intervention | 6 [3.5 to 7.5] | 4 [2 to 6]
Statistical Analysis 1: Comparison: Intervention vs Sham; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Isometric Maximum Voluntary Contraction (IMCV) in Newton (N) Right Knee-extensor
Description: It will be evaluated by isometric MCV (Newton) at 90 degree angle in the knee joint.
Time Frame: after 4 weeks
Measure: Median (Inter-Quartile Range); unit: Newton
Arm/Group | Intervention | Sham
Number analyzed (Participants) | 13 | 11
Newton
  Pre-intervention | 115.1 [79 to 183] | 141.4 [95 to 143]
  Post-intervention | 127.1 [93 to 164] | 128.7 [69 to 172]
Statistical Analysis 1: Comparison: Intervention vs Sham; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Ismometric Maximal Voluntary Contraction (IMVC) Left Knee-extension
Description: It will be evaluated by isometric MCV (Newton) at 90 degree angle in the knee joint.
Time Frame: after 4 weeks
Measure: Median (Inter-Quartile Range); unit: Newton
Arm/Group | Intervention | Sham
Number analyzed (Participants) | 13 | 11
Newton
  Pre-intervention | 83.2 [68 to 195] | 115.8 [77 to 176]
  Post-intervention | 154 [91 to 211] | 129 [48 to 166]
Statistical Analysis 1: Comparison: Intervention vs Sham; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Isometric Rate of Force Development (IRFD) Right Knee-extensor
Description: It will be evaluated by isometric RFD (Newton/seconds) at 90 degree angle in the knee joint.
Time Frame: after 4 weeks
Measure: Median (Inter-Quartile Range); unit: Newton/seconds
Arm/Group | Intervention | Sham
Number analyzed (Participants) | 13 | 11
Newton/seconds
  Pre-intervention | 489.8 [223 to 1307] | 558.5 [412 to 1272]
  Post-intervention | 510 [295 to 1166] | 560 [256 to 906]
Statistical Analysis 1: Comparison: Intervention vs Sham; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Isometric Rate of Force Development (IRFD) Left Knee-extensor
Description: It will be evaluated by isometric RFD (Newton/seconds) at 90 degree angle in the knee joint.
Time Frame: after 4 weeks
Measure: Median (Inter-Quartile Range); unit: Newton/seconds
Arm/Group | Intervention | Sham
Number analyzed (Participants) | 13 | 11
Newton/seconds
  Pre-intervention | 284.7 [190 to 1100] | 546.2 [347 to 920]
  Post-intervention | 580.3 [247 to 1140] | 521 [154 to 793]
Statistical Analysis 1: Comparison: Intervention vs Sham; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: zero period
Arm/Group | Intervention | Sham
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/11
Other Adverse Events (participants affected / at risk) | 0/13 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No